CLINICAL TRIAL: NCT03427918
Title: The Effectiveness of the Mindfulness-based Cognitive Therapy (MBCT) on Sexual Functioning in Epileptic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir H Pakpour, Director of Social Determinants of Health Research Center (SDH), Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1396.169
Record Dates: First submitted 2017-12-09; First posted 2018-02-09 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Epilepsy; Sexual Dysfunction
MeSH Terms: conditions — Epilepsy; Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patient-partner (Experimental): patients and their partners will receive a weekly Mindfulness-Based Sex Therapy program. The treatments will deliver by a group of facilitators to groups of women consisting of 4-7 women.
  Interventions: Behavioral: Mindfulness-Based Sex Therapy
- patient-partner and health care providers (Experimental): patients and their partners as well as health care providers will receive a weekly Mindfulness-Based Sex Therapy program. Th treatments will deliver by a group of facilitators to groups of women consisting of 4-7 women.
  Interventions: Behavioral: Mindfulness-Based Sex Therapy
- Control group (No Intervention): The control group will receive a routine counseling

INTERVENTIONS:
Behavioral: Mindfulness-Based Sex Therapy — Mindfulness-Based Sex Therapy in an integration of psychoeducation, sex therapy, and mindfulness-based skills.
  Arms: patient-partner; patient-partner and health care providers

SUMMARY:
Female sexual dysfunction (FSD) includes impairments in sexual desire, arousal, orgasm, and genital pain resulting in significant subjective distress. This study is aimed to assess a mindfulness-based intervention for improving sexual functioning among women with epilepsy

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Female sexual dysfunctions are categorized by the DSM-5 as sexual interest/arousal disorder, genitopelvic pain/penetration disorder, and female orgasmic disorder. The diagnoses require symptoms to be present for six months or more,
* Currently in a relationship that has lasted longer than 1 year
* Both members of the couple are able to speak and read Persian
* Both members of the couple provide signed and dated informed consent form

Exclusion Criteria:

* Cognitive impairment or mental illness that would impair ability to provide consent or participate in the program
* Major psychiatric disorder (e.g., psychosis, personality disorder)
* Current suicidal ideation or suicide attempt within past 3 months
* Past participation in an MBCT program

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 660 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Sexual functioning | changes from baseline, 1 Months and 6 months
  Sexual functioning is assessed using self-reported measure , female Sexual Function Index (FSFI)
Intimacy | changes from baseline, 1 Months and 6 months
  Personal Assessment of Intimacy in Relationships (PAIR) will use to assess relationship satisfaction. The PAIR is a self-reported measure with 36 items which cover five subscales
sexuality-related distress | changes from baseline, 1 Months and 6 months
  The Female Sexual Distress Scale revised version (FSDS-R) is extensively validated and among the most widely used tools to measure sexually related personal distress.

SECONDARY OUTCOMES:
Mindfulness for sexual functioning | changes from baseline, 1 Months and 6 months
  Sexual Five-Facet Mindfulness Questionnaire (FFMQ-S) is used to assess mindfulness in the context of sexual encounters.
Marital satisfaction | changes from baseline, 1 Months and 6 months
  The Maudsley Marital Questionnaire (MMQ) is a 20-item instrument measuring marital satisfaction.
Psychological distress | changes from baseline, 1 Months and 6 months
  Hospital Anxiety and Depression Scale (HADS) is a brief self-administrated tool to assess psychological distress in patients as well as general populations
Erectile Function | changes from baseline, 1 Months and 6 months
  International Index of Erectile Function Questionnaire (IIEF) is a self-reported and multidimensional measure of male's sexual function
quality of life | changes of QOLIE-31-P from baseline, 1 Months and 6 months
  QOLIE-31-P will be used to assess patient's quality of life

CONTACTS AND LOCATIONS:
Locations (15):
- Iran (15):
  - Abbasi, Karaj
  - Brain and Neuropsychological Clinic, Karaj
  - Shahid Madani, Karaj
  - Shahid Rejaei, Karaj
  - Mehregan, Qazvin
  - Razi Hospital, Qazvin
  - Attar clinic, Tehran
  - Baharlu Hospital, Tehran
  - Lolagar Hospital, Tehran
  - Raha, Tehran
  - Rasoul Akram Hospital, Tehran
  - Rezaei Clinic, Tehran
  - Sadaf, Tehran
  - Sina, Tehran
  - Ziaeian, Tehran

IPD SHARING:
Plan to Share IPD: Undecided